CLINICAL TRIAL: NCT05640427
Title: Effect of Different Doses of Dexmedetomidine on Cerebral Oxygen Saturation and Postoperative Anxiety in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022ZH0218
Record Dates: First submitted 2022-11-26; First posted 2022-12-07 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2022-12

CONDITIONS: Anxiety
Keywords: Dexmedetomidine; Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Placebo Comparator): Group C received general anesthesia with intravenous normal saline. The cognitive function of this groups was assessed with the Mini Mental State Scale (MMSE) on the day before surgery. the anxiety of this groups was assessed with Self-rating Anxiety Scale (SAS) on the day before, one day after and three days after surgery.
  Interventions: Drug: normal saline
- Group D1 (Experimental): groups D1 received general anesthesia with intravenous pump of 0. 2μg/kg/h dexmedetomidine. The cognitive function of this groups was assessed with the Mini Mental State Scale (MMSE) on the day before surgery. the anxiety of this groups was assessed with Self-rating Anxiety Scale (SAS) on the day before, one day after and three days after surgery.
  Interventions: Drug: Dexmedetomidine
- Group D2 (Experimental): groups D2 received general anesthesia with intravenous pump of 0. 5μg/kg/h dexmedetomidine. The cognitive function of this groups was assessed with the Mini Mental State Scale (MMSE) on the day before surgery. the anxiety of this groups was assessed with Self-rating Anxiety Scale (SAS) on the day before, one day after and three days after surgery.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Groups D1 received general anesthesia with intravenous pump of 0. 2μg/kg/h dexmedetomidine to 30min before the end of the operation.Groups D2 received general anesthesia with intravenous pump of 0. 5μg/kg/h dexmedetomidine to 30min before the end of the operation.
  Arms: Group D1; Group D2
Drug: normal saline — The same capacity of 0.9% normal saline was used in group C
  Arms: Group C

SUMMARY:
To investigate the effect of different doses of dexmedetomidine on Cerebral Oxygen Saturation and Postoperative anxiety in elderly patients undergoing laparoscopic surgery

DETAILED DESCRIPTION:
A total of 105 patients who were admitted to The First Hospital of Qinhuangdao for laparoscopic surgery and divided into control group (group C), dexmedetomidine doses of 0.2 μg/kg (group D1), dexmedetomidine doses of 0.5 μg/kg (group D2).

105 patients were randomized equally into 3 groups. 35 cases in each group. Group C received general anesthesia without dexmedetomidine, groups D1 received general anesthesia with intravenous pump of 0. 2μg/kg/h dexmedetomidine, groups D2 received general anesthesia with intravenous pump of 0. 5μg/kg/h dexmedetomidine.SBP(Systolic Blood Pressure),DP(Diastolic Pressure),HR(Heart Rate) and rScO2(Regional cerebral oxygen saturation) of the three groups were recorded before anesthesia induction (T1), at the time of intubation (T2), five minutes after induction(T3),at the beginning of surgery (T4), immediately after surgery (T5), and five minutes after extubation (T6).

The cognitive function of the three groups was assessed with the Mini Mental State Scale (MMSE) on the day before surgery. the anxiety of the three groups was assessed with Self-rating Anxiety Scale (SAS) on the day before surgery,one day after and three days after surgery, comparing the incidence of anxiety between the three groups. Analyze whether dexmedetomidine reduced the incidence of anxiety by increasing cerebral oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years or older who underwent elective laparoscopic surgery under general anesthesia
* BMI less than 30 kg/m2
* American Society of Anesthesiologists (ASA) grades I-III
* The score of Mini Mental state examination≥24

Exclusion Criteria:

* Patients with heart, lung and other vital organ disorders
* The score of Mini Mental state examination≤23
* Preoperative psychiatric disorders or long-term use of drugs affecting the psychiatric system
* Have severe visual, hearing, speech impairment or other inability to communicate with the visitor
* Refuse to sign informed consent
* known preoperative left ventricular ejection fraction less than 30%, sick sinus syndrome, severe sinus bradycardia (<50 beats per min [bpm]), or second-degree or greater atrioventricular block without pacemaker

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Incidence of anxiety at one day after surgery | One day after surgery
  The three groups of patients were scored on the Self-rating Anxiety Scale on the first day after surgery, and if the Self-rating Anxiety Scale score was ≥ 50 points, the patients developed anxiety, and whether the incidence of anxiety on the first day after surgery in the three groups was statistically significant.
Incidence of anxiety at three days after surgery | Three days after surgery
  The three groups of patients were scored on the Self-rating Anxiety Scale on the third day after surgery, and if the Self-rating Anxiety Scale score was ≥ 50 points, the patients developed anxiety, and whether the incidence of anxiety on the third day after surgery in the three groups was statistically significant.

SECONDARY OUTCOMES:
Anesthetic drug | Time Frame: during the surgery
  The dosage of remifentanil and propofol in different groups were recorded.
The change of SBP | before anesthesia induction, at the time of intubation, at the beginning of surgery, immediately after surgery , and five minutes after extubation
  The change of Systolic blood pressure (SBP) among the three groups.
The change of rScO2 | during the surgery
  The change of regional cerebral oxygen saturation(rScO2) among the three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Shujuan Liang, Master, Study Director — The First hosptial of Qinhuangdao; Hua Zhou, Master, Study Chair — The First hosptial of Qinhuangdao
Locations (1):
- The First hosptial of Qinhuangdao, Qinhuangdao, Hebei, China

IPD SHARING:
Plan to Share IPD: No